CLINICAL TRIAL: NCT04721301
Title: LUMINESCENCE-001 Ipilimumab, Maraviroc and Nivolumab in Advanced Metastatic Colorectal and Pancreatic Cancer
Brief Title: Ipilimumab, Maraviroc and Nivolumab in Advanced Metastatic Colorectal and Pancreatic Cancer the LUMINESCENCE Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: German Cancer Research Center (Other)
Responsible Party: Principal Investigator, Niels Halama, Principal Investigator, Head of Department Translational Immunotherapy, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-003297-13
Record Dates: First submitted 2020-11-12; First posted 2021-01-22 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer Metastatic; Pancreatic Cancer Metastatic
Keywords: microsatellite stable; immunotherapy
MeSH Terms: interventions — Nivolumab; Ipilimumab; Maraviroc

STUDY DESIGN:
Intervention Model Description: Single Center Phase 1 trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination immunotherapy (Experimental): Treatment arm with Nivolumab, Ipilimumab and Maraviroc combination treatment
  Interventions: Combination Product: Nivolumab plus Ipilimumab plus Maraviroc

INTERVENTIONS:
Combination Product: Nivolumab plus Ipilimumab plus Maraviroc — In the single treatment arm, all patients receive Nivolumab, Ipilimumab and Maraviroc

SUMMARY:
The study will be conducted in compliance with Good Clinical Practices (ICH-GCP) and the Declaration of Helsinki, and in accordance with applicable legal and regulatory requirements, including archiving of essential documents.

DETAILED DESCRIPTION:
A study to evaluate the safety, tolerability and feasibility of treatment with Maraviroc, nivolumab and ipilimumab in layers of colon and pancreatic cancer patients

ELIGIBILITY:
Inclusion Criteria:

* written informed consent given, signed and dated
* age ≥ 18 years
* male or female patient with a history of treated metastatic stage IV colorectal or pancreatic cancer with liver metastases of the primary colorectal or pancreatic cancer
* histologically confirmed primary colorectal or pancreatic cancer
* preferentially with metastatic lesion in the liver amenable to biopsy (must have at least one measurable lesion or evaluable disease by CT or MRI per RECIST criteria measured within 56 days prior to trial inclusion)
* expected survival of at least three months
* Karnofsky performance status > 70 %
* patients that have received current standard treatment options (or could not receive treatment due to medical reasons, e.g. allergic reactions, contraindications, toxicities etc.) for colorectal cancer (oxaliplatin or irinotecan in combination or alone with 5-FU with or without treatment combinations of cetuximab and/or bevacizumab or panitumumab, trifluridine plus tipiracil) or patients with pancreatic cancer that have received standard treatment options (at least first line therapy, progression or intolerance to oxaliplatin, irinotecan and 5-FU, FOLFIRINOX as first or second line therapy) or platinum containing adjuvant chemotherapy and palliative after first line chemotherapy
* no chemotherapy treatment within the last two weeks (to baseline)
* within the last 2 weeks prior to study day 1 the following laboratory parameters, which should be within the ranges specified:

Laboratory Parameter Range Absolute neutrophil count (ANC) ≥ 1000/mm3 (≥ 1.0 x 109/L) Platelets ≥ 50.000/mm3 (≥ 80 x 109/L) Creatinine Clearance limit as assessed by GFR > 360 mL/min/1.73m² ALT and AST < 3.0 x ULN (w. liver met.) total bilirubin hemoglobin < 1.5 x ULN >9 g/dl

* ability to understand character and individual consequences of the clinical trial
* if the patient is female, she must be of non-childbearing potential, or practice highly effective contraception (Pearl Index <1%, e.g. intrauterine device (IUD)) while receiving study drug and up to 5 months from the last dose of study drug.
* if the patient is male, he must continue contraception for at least 31 weeks (90 days plus the time required for nivolumab to undergo 5 half-lives) after the last dose of investigational drug. In addition, male patients must abstain from sperm donation during this time

Exclusion Criteria:

Patients presenting with any of the following criteria will not be included in the trial:

* Patients with severe kidney disorders (GFR of <30 mL/min/1.73m² and diagnosed kidney disease) or who are on hemodialysis.
* The patient requires concomitant chronic treatment with systemic corticosteroids or any other systemic immunosuppressive agents. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease (See also Section 7.7)
* Patients taking immunomodulatory medication (e.g. Type 1 interferons).
* Current use of any investigational or non-registered product (drug or vaccine) other than the study treatment
* Patients with a single metastatic lesion without identified concomitant lymph node metastasis (i.e. a patient with the intent to resect the metastasis)
* Patients with metastatic colorectal or pancreatic cancer that have a drastic clinical progression (e.g. from Karnofsky performance 100% to 70%) within the last six weeks before screening cannot participate
* The patient with active autoimmune disease or with a history of autoimmune disease.
* The patient has a family history of congenital or hereditary immunodeficiency.
* The patient is known to be positive for Human Immunodeficiency Virus (HIV) or other chronic infections (HBV, HCV) or has another confirmed or suspected immunosuppressive or immunodeficient condition.
* The patient has concurrent chronic severe medical problems (significant heart failure, uncontrolled diabetes, bleeding disorder, interstitial lung disease, etc.), unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
* Patients with untreated known CNS metastases, patients are eligible if CNS metastases are adequately treated and patients are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to trial participation.
* The patient has previous or concomitant malignancies at other sites, except effectively treated carcinoma in situ of the cervix or effectively treated malignancy that has been in remission for over 5 years and is highly likely to have been cured.
* For female patients: the patient is pregnant or lactating.
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product
* Known allergy or hypersensitivity to peanuts, soy, soy beans or derivatives of soy or peanuts
* Contra-indication for MRI
* Participation in another clinical trial within three weeks before screening day
* Patient will not be allowed to enroll in this trial more than once.
* Known microsatellite-instability (MSI-H or dMMR) as evidenced by a standard laboratory practice (e.g. PCR or staining or sequencing etc.)
* Prisoners or patients who are involuntarily incarcerated.
* Patients who are compulsorily detained for treatment of either a psychiatric or physical(e.g., infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Number of participants and severity of treatment-related adverse Events as assessed by CTCAE v4.0 | up to 11 days
  Safety and tolerability of combined Maraviroc, Ipilimumab and Nivolumab

SECONDARY OUTCOMES:
Progression Free Survival | up to 36 months
  Progression free survival after initiation of trial medication, time to progression on trial medication, radiologic evaluation based on RECIST and iRECIST criteria
Overall Survival | up to 36 months
  Overall survival after initiation of trial medication, radiologic evaluation based on RECIST and iRECIST criteria
Tissue Response | up to 3 months
  Detailed evaluation of in-treatment biopsy compared to pre-treatment biopsies, investigating overt tumor cell death, immune cell activation, immune cell density and general markers of proliferation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Heidelberg / NCT, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided